CLINICAL TRIAL: NCT07336407
Title: Data Collection for the Validation of an AI Software to Support MSK Ultrasound Examination
Brief Title: Data Collection for the Validation of an Artificial Intelligence Software to Support Musculoskeletal Ultrasound Examination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Smart Alfa Teknoloji San. ve Tic. A.S. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MSK-001-02
Record Dates: First submitted 2026-01-11; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Ultrasound Imaging of Anatomical Structures
Keywords: Musculoskeletal; Artificial Intelligence; ultrasound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- U.S population (Other)
  Interventions: Device: Ultrasound Scans

INTERVENTIONS:
Device: Ultrasound Scans — Scanning for musculoskeletal examination views on shoulder, elbow, wrist/hand, knee, and foot/ankle.

SUMMARY:
This study conducted at three locations, aiming to collect ultrasound images from volunteers and assess the performance of an AI software, MSK Go, using these images.

The software to be assessed is designed to assist physicians and healthcare professionals in performing ultrasound exams by classifying scan views and identifying key anatomical structures during a musculoskeletal ultrasound examination.

The main question the study aims to answer is whether the AI software performs safely and effectively for future clinical use.

DETAILED DESCRIPTION:
This study is designed to validate the performance of the MSK Go software in classifying musculoskeletal ultrasound examination views and segmenting relevant anatomical structures in a U.S. population.

Data collection method and analysis:

A total of 79 subjects were enrolled and undergone shoulder, elbow, wrist/hand, knee, and foot/ankle scans at three clinical sites. Ultrasound examinations were performed by MSK ultrasound experts without using MSK Go.

Each participant spent approximately 30 minutes in the ultrasound scanning session. Demographic data were collected for all subjects. An FDA-cleared, commercially available ultrasound device was used at each location.

The collected ultrasound scans are then annotated by healthcare professionals with expertise in musculoskeletal sonography.

In a post hoc analysis, the ultrasound clips were processed using the AI software, and the software-generated classifications of views and segmentations of anatomical structures were compared with the reference annotations .

Convenience sampling was applied during data collection to ensure that participants represented a balanced distribution across age, gender, BMI, and ethnicity.

ELIGIBILITY:
Inclusion Criteria:

* Provision of a signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study

Exclusion Criteria:

* Pregnancy
* Inability to lie flat
* Open skin lesions or active infection at the scan site
* Anatomical deformity in the joints to be scanned

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Rate of spatial (area) overlap of anatomical structure areas on the ultrasound image | Up to 30 days from enrollment
  The performance based on the rate of the spatial (area) overlapping of supported structures
Rae of correctly classifying the views of the joint | Up to 30 days from enrollment
  The performance based on the rate of correctly detecting views of the selected joint

SECONDARY OUTCOMES:
Rate of correctly assigning anatomical structure completeness level for any scan view of the joint | Up to 30 days from enrollment
  The performance based on the completeness rate of detection level of the set of supported anatomical structures by the software

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Scripps Clinic Torrey Pines, La Jolla, California
  - AABP Integrative Pain Care and Wellness Clinic, Brooklyn, New York
  - Memorial Hermann Houston Health & Sports Medicine, Woodland, Texas

IPD SHARING:
Plan to Share IPD: No